CLINICAL TRIAL: NCT03416686
Title: Radiofrequency in Differentiated Thyroid Cancer Metastatic Lymph Node: Prospective Study of Safety and Efficacy
Acronym: METATHYRAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P170201J
Record Dates: First submitted 2017-12-07; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Differentiated Thyroid Cancer
Keywords: differentiated thyroid cancer; Radiofrequency

STUDY DESIGN:
Intervention Model Description: Radiofrequency with local anesthesia: 1 episode of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency (Experimental)
  Interventions: Device: Radiofrequency (RF star electrode electrode_Fixed)

INTERVENTIONS:
Device: Radiofrequency (RF star electrode electrode_Fixed) — The radiofrequency will be performed under ultrasound control after local anesthesia by a trained operator, after finding the lesion to be treated by the operator.
  Medical device used: RF star electrode electrode_Fixed (Starmed Co,Gyeonggi-do, Korea, French representative Cosysmed).

SUMMARY:
Radiofrequency (RF) could be technically feasible and effective in the treatment of lymph node metastases of differentiated thyroid cancer. It could constitute a minimally invasive and feasible therapeutic alternative in ambulatory, allowing a reduction of the tumoral volume sufficient to limit the symptoms even to induce a tumor remission, a normalization of the tumoral markers and a better quality of life.

The aim of this study is to evaluate the anti-tumor echographic efficacy at 12 months of radiofrequency on lymph node (LN) metastasis of thyroid cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients over age of 18 years
* with differentiated thyroid cancer (papillary, follicular) histologically confirmed, and absence of anaplastic component
* Previous treatment by total thyroidectomy and cervical lymph node dissection.
* Previous treatment by at least 1 therapeutic radioactive iodine (minimum activity 740MBq)
* Persistence on cervical ultrasound of at least 1 cervical metastatic lymph node, visible at ultrasound, small diameter between ≥10 mm and ≤30mm, volume maximum 20ml, spotted on a picture, and confirmed by cyto-punction
* Signed informed consent

Exclusion Criteria:

* Location of LN metastasis with significant risk of local complication (nervous, vascular) according baseline ultrasound assessment
* Patient carrier of a pacemaker or a defibrillator
* Congenital or acquired hemostasis abnormality, anticoagulant therapy or double platelet antiaggregatory (aspirin and clopidogrel)
* Hypersensitivity to local anesthetic
* Poor general condition (performance status Eastern Cooperative Oncology Group (ECOG) > 1)
* Survival estimated less than 12 months
* Patient who can't follow the instructions of RF therapy or who can't be followed during 2 years in order to meet the objectives of the study
* Non affiliation to a social security
* Pregnant or breast feeding women at the time of RF
* Beta hormone chorionic gonadotrope (HCG) positive test (pregnancy) before RF therapy
* Baseline cervical ultrasound, by expert operator trained to RF, not fulfilling feasibility criteria for RF realisation because of the location of LN metastasis or the way to reach it
* Controlateral recurrent palsy on nasofibroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Treatment response. | 12 months
  Treatment success wil; be defined on the following three criteria that should be all fulfilled
  * Loss of metastatic aspect on ultrasonography
  * LN decreased volume at least 50%
  * no vascularization in Doppler

SECONDARY OUTCOMES:
Percentage of patients with non-suspicious cyto-punction of treated LN at 6 months after RF | 6 months
Percentage of patients without any new suspicious cervical lesion | 3, 6, 12 and 24 months.
Response time | within 38 months
  response time for partial response, major response and disappearance of lymph node at ultrasound.
Reduction in thyroglobulin level in blood | 3, 6, 12 and 24 months
Reduction in thyroglobulin antibody level in blood | 3, 6, 12 and 24 months
Percentage of patient in tumor response | 12 and 24 months
  Tumor response is defined according American Thyroid Association's criteria
Percentage of patients without any new therapeutic event | 12 and 24 months
Percentage of patients with good immediate tolerance | day 0
Percentage of (either expected or unexpected) clinical complications | 3, 6, 12 and 24 months
Percentage of patients who had a RF complete procedure | day 0
Percentage of patients who had a RF incomplete procedure | day 0
Anxiety | 3, 6, 12 and 24 months
  visual analog scale coted by the patient
36-item Medical Outcomes Study Short-Form Health Survey (SF-36) | 3, 6, 12 and 24 months
  it measures the quality of life
EuroQol (EQ-5D) | 3, 6, 12 and 24 months
  EQ-5D is a standardized instrument for measuring generic health status. Health status is measured in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided